CLINICAL TRIAL: NCT06920940
Title: Child Bipolar Network Ketogenic Diet Approach to Bipolar Disorder in Adolescents
Acronym: CBN Keto
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of Cincinnati (Other); University of Pittsburgh (Other); University of Colorado, Denver (Other); Advanced Ketogenic Therapies (Unknown); Baszucki Family Foundation (Unknown)
Responsible Party: Principal Investigator, David J. Miklowitz, Ph.D., Distinguished Professor of Psychiatry, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB#24-5711
Record Dates: First submitted 2025-03-26; First posted 2025-04-10 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-03

CONDITIONS: Bipolar Disorder (BD); Bipolar Disorder NOS; Bipolar Disorder I or II; Bipolar Spectrum Disorder; Adolescents
Keywords: ketogenic; treatment; diet; keto
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ketogenic Therapy for Bipolar Spectrum Disorders (Experimental): This is a pilot trial with one intervention arm. All youth meeting eligibility for the ketogenic therapy phase of this pilot trial will be invited to participate in the intervention and progress tracking.
  Interventions: Other: Ketogenic Therapy

INTERVENTIONS:
Other: Ketogenic Therapy — During the keto therapy (16 weeks), the youth will participate in a strict ketogenic diet, with adjustments made as necessary from weekly dietitian coaching sessions.

SUMMARY:
The present study is an open trial of ketogenic diets for adolescents and young adults (ages 12-21 yrs) in the depressive or mixed phases of bipolar disorder (BD). The investigators aim to determine whether combining standard of care pharmacological treatment for bipolar spectrum disorders with a 16-week ketogenic diet is well-tolerated and associated with improvements in depression, inflammatory and metabolic indicators, and executive functioning over the study period.

The experimental treatment in this study is a 16-week full ketogenic diet. Four study sites (UCLA, U Cincinnati, U Colorado and U Pittsburgh) will recruit 80 total youth (20 each) from bipolar specialty clinics. All youth eligible for the ketogenic therapy will be provided with the ketogenic diet and standard of care pharmacological treatment. During the diet therapy youth will be seen by a study child/adolescent psychiatrist at least once a month (and more frequently when needed), with the psychiatrist recommending and providing side effects monitoring and pharmacotherapy as clinically indicated.

The youth and caregivers will also meet with an expert dietitian who will coach all youth on maintaining the ketogenic diet (low carbs, high fats, medium protein) and making sure the child is tolerating the diet and getting enough liquid and nutrients, following the practice guidelines of the International Ketogenic Diet Study Group for treating youth. All youth and involved caregivers will also be provided will at least one motivational enhancement session to support them in goal setting and completion of the study elements.

Throughout the study the investigators will assess metabolic (e.g., blood ketones, HOMA-IR) and inflammatory indicators (e.g., C-reactive protein), both for safety reasons and to assess correlates of symptomatic change. Independent evaluators will assess youth every month regarding their symptoms (depression, mania, anxiety, psychosis), psychosocial functioning, and quality of life.

The investigators anticipate that the pilot will transpire over 24 months and be an important step toward establishing feasibility and acceptability of ketogenic therapy for this population, not only in terms of diet administration and compliance but also for obtaining symptomatic, metabolic and inflammatory measurements.

DETAILED DESCRIPTION:
Site PIs David Miklowitz, Ph.D., Distinguished Professor of Psychiatry, University of California, Los Angeles

Danella Hafeman, M.D. and Boris Birmaher, MD, University of Pittsburgh School of Medicine;

Christopher Schneck MD (site PI), Melissa Batt, MD (co-PI), and Aimee Sullivan, PhD, University of Colorado Anschutz Medical Campus, Aurora, CO.

Melissa Delbello, MD (site PI) and L. Rodrigo Patino Duran, MD (Co-PI), University of Cincinnati College of Medicine

Phase 1: Intake Period and Pre-Treatment Assessments

During the approximately 4-week intake period (phase I) the investigators will conduct a psychiatric and medical evaluation of the child to determine whether the youth meets diagnostic, symptom, and keto trial eligibility and the diet is consistent with the youth's health goals.

Phase I: Evaluation Phase Steps

1. An initial phone screen will be completed with potential young adult participants, or one or more parents or legal guardians for potential minor participants. If they remain potentially eligible and interested, they will be invited to come to the clinic for the consenting process. If a minor has two parents or guardians with legal rights to health care decision making, both parents need to sign consents.
2. If youth and their parent(s) assent/consent, they will move on to phase 1 psychiatric evaluation (diagnostic interview, symptom assessment, psychiatric and medical history) with a study psychologist and psychiatrist
3. Families and youth will go to the UCLA Clinical and Translational Research Center (CTRC) for venipuncture and a urine sample. Blood draws will be performed by either certified phlebotomy technicians or registered nurses. Intake blood tests required prior to starting keto diets include lipids, insulin, glucose, thyroid-stimulating hormone test, A1C, and cholesterol (see Table 2 for a complete list); total blood volume to be collected at intake is a little less than 2 tablespoons)
4. Families and youth will next meet with the study dietitian (Denise Potter, RDN or her designee) who will (a) perform a separate assessment of the child's eligibility for the study, and (b) provide education about the diet (e.g., expected benefits and side effects, the importance of regular ketone assessments). Study clinicians (psychiatrists, psychologists, and dietitians) will jointly determine the youth's eligibility in term of diagnosis, symptom status, and health for initiation of keto therapy, which begins in phase II.
5. If youth is eligible for ketogenic therapy and decides to continue, they will be invited to continue and to next meet with a study therapist (e.g., psychologist, social worker, MH counselor) for (a) a 45-60 min family psychoeducation session concerning how to cope with BSDs (for example, how to recognize prodromal symptoms of mania and work with the treatment team to prevent recurrences) and the role of nutrition; and (b) a 45-min individual session for the youth ("motivational enhancement" sessions) to explore the youth's health-related goals, values, and motivation for initiating and completing the diet phase.

Following best practice guidelines for the treatment of bipolar disorder participants will be assigned a study psychiatrist with expertise in pediatric mood disorders for their initial medication consultation. During the 16-week keto trial, the psychiatrist will review lab and test results and meet with youth/parents at least monthly to oversee safety of medications prescribed. The psychiatrist will work to stabilize the youth on psychiatric medications prior to initiation of diet therapy in phase II. However, this is not a psychopharmacology study: youth are not required to start or stop any medications to participate in the keto phase (II) of the study. During the monthly visits, psychiatrists will help participants address any side effects or safety concerns, including making clinically necessary medication adjustments (e.g., increasing the dose of a mood stabilizer to treat depression). Psychiatrists will coordinate with the study's registered dietitian and other relevant care professionals (e.g., the youth's GP) as needed. This plan for psychiatrist care aligns with best practice guidelines for youth with BSDs.

Phase II: Ketogenic Preparation and "Ramp Up"

Once the youth and parents have consented to the study and been determined to be eligible for keto therapy, phase II will begin with a 2-3 week period of diet adjustment or "ramping up." During this 2-3 week period, they will meet with the dietitian weekly to discuss some simple keto recipes (e.g., for lunch) and problem-solve regarding barriers to implementing the diet. This period helps reduce the likelihood of side effects from the transition in diet (e.g., Keto flu) by easing the participant into the low carb state and getting them used to self-administered blood ketone assessments. This is accomplished, for example, by cutting out sugar and introducing a single self-prepared keto meal each day for one week, and then two keto meals in the second week, and three in the third. Prior to starting the official diet, participants will complete a pre-diet assessment of mood symptoms, psychosocial functioning, surveys, and brief neuropsychological testing. They will also take pictures of their meals and snacks for 3 days prior to phase III (to be uploaded to a HIPAA-compliant box folder and shared with the dietitian and study team). If the youth has adjusted well during the ramp up period, the diet therapy trial (phase III) will be initiated and the 16-week diet therapy clock will start.

Phase III. Keto Therapy Trial

During the keto therapy phase (16 weeks), the dietitian will help the family and youth order keto meals from Factor 75 (a food delivery service), with adjustments made as necessary from weekly dietitian coaching sessions. The prescribed keto diet aligns with practice guidelines of the International Ketogenic Diet Study Group for youth. The family may choose to buy their own groceries and cook their own keto meals for the youth rather than having the meals delivered, and if so they will be compensated for groceries on a per diem basis by the study. The dietitian will monitor the youth's dietary intake, baseline blood ketone and lipid/cholesterol/insulin/glucose values, and potential dietary side effects at weekly visits. The youth be asked to take a daily self-administered blood test (fingerprick) using a "Keto Mojo" meter provided to them, which will tabulate level of ketones and glucose. These readings will be entered into a HIPAA-compliant server and accessed by the study dietitian and research team. The repeat readings will help determine whether the youth achieves and maintains a state of ketosis, which is the goal of ketogenic diets.

The youth will return to the CTRC lab for a repeat blood test (glucose, lipids, inflammatory markers, etc.; see Table 2 for complete list of tests) at 8 weeks (mid-treatment) and 16 weeks (end of study) so that the dietitian and psychiatrist can track the youth's health and response to the diet. Independent evaluators will interview participants every 4 weeks through the 16-week study for symptoms (e.g., depression, mania, anxiety, mood instability) and psychosocial functioning.

Phase IV: Post-Treatment Assessments

At the end of the 16-week keto trial, a post-treatment evaluation will be conducted with the same measures (symptom assessments, neuropsychological functioning, psychosocial functioning) done at intake. Participants will be compensated for completing all research measures.

Specific Aims

Hypothesis #1: Diet Adherence and Tolerance. An estimated 60 youth (15 per site) in bipolar depressed or mixed states (depressed with hypomanic or manic symptoms) will be cleared for initiation of the 16-week keto diet following an initial 4-6-week intake assessment and preparation period. The investigators expect 40 (10 per site) to complete the 16-week keto therapy trial and post-assessment. The investigators will assess the proportion of youth who maintain ketosis, as measured through (a) daily blood ketone assays using the Keto Mojo device, a Bluetooth-enabled ketone and glucose testing kit, and (b) photographs of food intake (meals, drinks, and snacks) one day per week. The investigators will assess diet tolerance and safety through calculating the proportion of youth staying on the diet, parent and youth reports of side effects, and dietitian- and independent evaluator-collected side effect questionnaires. The investigators hypothesize that with appropriate coaching, the investigators will observe keto diet compliance rates of 70-80%. The investigators hypothesize that the diet will be sufficiently tolerated, with family participants and clinicians reporting that side effects are manageable.

Hypothesis #2: Symptom Improvement. Youth with high compliance to the 16-week keto diet will have significant reductions in bipolar depressive symptoms from baseline to completion of the 16-week diet, without concomitant increases in hypomanic symptoms. The investigators further expect that they will show significant reductions in mood instability and increases in Global Assessment of Functioning scores (rated on a 1-100 scale).

Hypothesis #3. Metabolic Indicators. Youth with high compliance with the keto diet will show significant pre- to post-treatment improvement in metabolic indicators (e.g., insulin resistance and glucose values (HOMA-IR), inflammatory markers (e.g., CRP), and cognitive (executive) functioning from baseline to end of treatment.

Background and Significance

Bipolar spectrum disorders (BSDs) affect approximately 2.5% of children and adolescents worldwide. Youth with BSDs are at high risk for recurrent courses of illness and poor psychosocial functioning even when receiving pharmacotherapy. When treated with standard mood stabilizers or antipsychotics, only 43% of adolescents with bipolar I disorder recover in the year after a hospitalized manic episode; 54% have illness recurrences and as many as 1 in 3 are treatment refractory. Moreover, only 35% are adherent with prescribed medications during the post-hospital year. The investigators need more effective and better-tolerated interventions for youth with bipolar I or II disorder, as well as those on the bipolar spectrum who are at risk for developing a full-blown bipolar I or II disorder (i.e., other specified bipolar disorder, with major depressive episodes alternating with recurrent periods of subthreshold mania or hypomania). The goals of early intervention for BSD are to fully stabilize youth from existing depressive episodes, prevent recurrences, and enhance individual functioning.

Depression is the primary unmet concern of most patients with BSD, regardless of age. Adult and youth patients with bipolar I or II spend three times as many weeks in their lives in depressive episodes compared to manic or hypomanic episodes. Undertreated depression is the strongest predictor of cognitive, metabolic and functional impairments associated with the disorder, including suicidal thoughts/behaviors, attention and memory impairments; and academic, occupational or social disability. Manic, mixed (depressive and hypomanic/manic), and hypomanic symptoms and episodes are also highly disruptive and impairing to youth. Most antipsychotic and mood-stabilizing agents are more effective in treating manic episodes than depressive or mixed presentations but are also associated with metabolic side effects such as weight gain and obesity. Clearly, the investigators need more effective treatments for bipolar depression and mixed phase (depressive and hypomanic/manic) presentations in youth.

What Can Be Done? Youth with BSD are usually treated with lithium, lamotrigine or second- generation antipsychotic agents (SGAs) such as lurasidone (Latuda) or aripiprazole (Abilify). All SGAs are associated with metabolic side effects, although some (e.g., lurasidone) cause fewer metabolic side effects than others (e.g., olanzapine). In the first two years of the Child and Adolescent Bipolar Network (CABIN) study (IRB-22-0309), the investigators implemented systematic pharmacological algorithms for the choice of primary and secondary agents, adjusting dosages, combining agents, and using adjunctive treatments to address side effects (for example, Metformin) in youth with bipolar depression or hypo/mania. In the CABIN study, there was substantial agreement among expert psychiatrists as to what medications were first and second-line choices for bipolar depression, mania, and mixed phases, whether bipolar I, II, or other specified in subtype. Nonetheless, it is clear to us from this and many other studies that a large proportion of youth with BSDs do not respond adequately to evidence-based medications alone.

Youth with or at risk for BSD are likely to have a long treatment course ahead of them and challenges with recovery. Testing whether ketogenic therapy - given adjunctively to pharmacotherapy - can help stabilize depressive or mixed symptoms and enhance cognitive and metabolic functioning in youth with BSD is of significant public health importance. To test the efficacy of keto therapy combined with pharmacotherapy, the investigators need to start with an open trial to test tolerability, feasibility, and adherence rates, and to determine whether there are clinical benefits that warrant evaluation in a randomized controlled trial.

Diet and Nutrition What is the role of diet and nutrition in the effort to stabilize mood episodes in bipolar youth? There is growing evidence that ketogenic diets are associated with mood improvement in adult bipolar patients and reductions in seizures in children with treatment- refractory epilepsy. As in epilepsy, BSDs are associated with neuroinflammation and oxidative stress. The ketogenic diet operates through strengthening antioxidant defenses, improving mitochondrial function, and regulating inflammatory genes.

There is increasing evidence that ketogenic diets are associated with improvements in executive functioning in elderly patients - enhanced working memory, planning ability, mental flexibility, and self-control. Executive functioning is impaired in bipolar disorder and is often in evidence even when individuals are not in a mood episode. Whether ketogenic diets improve executive functioning in psychiatric patients has not been adequately tested.

Importantly, ketogenic or other nutrition plans have never been tested systematically in youth with BSDs. This study provides a unique opportunity to test the mood- stabilizing effects of adjunctive ketogenic therapy and identify which subgroups of bipolar youth respond optimally to it. The investigators hypothesize that in a 16-week open trial youth with bipolar disorder will show substantial mood improvement on the combination of standard of care pharmacotherapy and ketogenic diets. In secondary analyses, the investigators will explore whether diet adherence (e.g., days in ketosis, as indicated by daily blood ketosis values and estimates of grams of carbohydrates consumed) is correlated with levels of improvement in mood and cognitive functioning over 16 weeks.

Youth with BSDs tend to have more impairment in metabolic indices such as BMI than their age-mates. Teens with impaired metabolic functioning are also likely to have poorer executive functioning. Although weight loss is not the purpose of keto therapy, t is possible that in early-onset BD, the subgroup of youths with impaired metabolic functioning will show the most symptom benefit and cognitive improvement with ketogenic diets. Indeed, a 12-week study in overweight teens found that a high fat, low-carbohydrate diet was associated with greater weight loss than a low-fat diet, and more improvement in HDL-C and triglyceride levels. In secondary analyses the investigators will explore the effects of a ketogenic diet on BMI and executive functioning over 16 weeks.

Research Design and Methods: Study Stages

This study is divided into four stages as follows, with more details on the steps and responsible staff noted in Table 1:

Phase I (~4 weeks total): the intake phase, where the potential participant is screened by telephone, consented for the study, and administered a battery of diagnostic and biological assays to determine study-eligibility.

Phase II (2-3 weeks total): the pre-keto preparatory phase, in which the youth will "ramp up" to the full 3 meal/day keto program by eating one keto meal per day in the first week, two in the second, and 3 in the third. The youth will also complete a pretreatment battery of symptom, functioning, and neuropsychological measures at this phase (interviews and self-report surveys).

Phase III (16 weeks total): the keto therapy trial.

Phase IV (1 week): the closing assessment and feedback phase.

ELIGIBILITY:
Inclusion Criteria:

* Youth must be ages 12 to 21 years old and speak English
* Youth must be appropriate for outpatient treatment (i.e., not a danger to self or others; not acutely psychotic, suicidal or manic; not in need of partial or full hospitalization)
* Youth must have a current BSD (bipolar I, II per DSM-5 criteria (Association, 2013) or other specified BSD by the University of Pittsburgh diagnostic criteria (Birmaher et al., 2006). The Pittsburgh other specified BSD criteria require recurrent and distinct 1-3 day periods (minimum 4 hours/day) in which there has been abnormally elevated, expansive, or irritable mood plus two (three, if irritable mood only) symptoms of mania that caused a change in functioning and totaled at least 4 days in the child's lifetime
* Active symptoms: In the 2 weeks prior to study intake, participants must have had weekly depression Psychiatric Status Ratings (PSRs) of 3 (moderate) or higher (using the 1-6 depression severity scales from the Adolescent Longitudinal Follow-up Evaluation, or A-LIFE); or an interview-based Children's Depression Rating Scale, Revised (CDRS-R) score covering the prior 2 weeks of > 20. Youth may also enter with mixed symptoms (e.g., simultaneous elevations of > 3 on the PSR depression and hypomania scales, with Young Mania Rating Scale scores of 12 or higher), without meeting criteria for a full manic episode in the past month.
* Participants must continue to meet the study's active symptom criteria when beginning the phase II keto "ramp-up" phase: a depression PSR rating of 3 or higher over the prior 2 weeks, and a CDRS-R score covering the prior 2 weeks of > 20.
* Youth/parents must be willing to participate in evaluation and medication management sessions with a study psychiatrist and the study dietitian for assessment of the diet and side effects.
* Youth under 18 years old must have at least one English-speaking parent or other caregiving family member consenting to participate in the study and available for consultation if needed
* Youth and (for minors) all parents/legal guardians with health care decision making rights must express willingness to have the youth be in the study and try the keto therapy, assuming that the youth is eligible. The team must ascertain that the participating minor's youth/caregiver is likely to make a strong effort to adhere to the study's protocol.

Exclusion Criteria:

The youth must not have any of the following needs or conditions for which the keto diet may be contraindicated:

* pregnancy or breastfeeding
* underweight (BMI below 18.5) or wasting syndrome (e.g., anorexia cachexia)
* current or history of anorexia nervosa
* current disordered eating (bulimia or binge eating disorder)
* autism spectrum disorder diagnosis level 2 or greater (more than mild)
* cardiac issues, including history of arrhythmia, or cardiovascular or cerebrovascular disease
* type I and type II diabetes
* history of seizures/epilepsy
* history of stroke or cancer
* unstable respiratory condition
* severe gastroesophageal reflux (GERD; painful/impairing despite prescription medication)
* substance use disorder (with an exception for mild cannabis or nicotine use disorders)
* history of kidney stones/disease
* diseases involving the pancreas, liver, gallbladder or thyroid, including Von Gierke's glycogen storage disease
* Condition with high cholesterol of triglycerides will prompt physician review of eligibility (LDL>190 or triglycerides>500)
* genetic metabolic disorders: either porphyria (impacting the body's ability to make hemoglobin) or fatty acid oxidation disorder (FAOD)
* rare conditions of defective ketone production or breakdown (carnitine deficiency, carnitine palmitoyl-transferase deficiency, carnitine-acylcarnitine translocase deficiency, mitochondrial fatty acid β-oxidation disorders, Succinyl-CoA:3-ketoacid CoA transferase deficiency (SCOT), or pyruvate carboxylase deficiency)
* youth must not be taking SGLT-2 inhibitors (e.g., canagliflozin), insulin, or sulfonylureas (to avoid hypogycemia), or Antihypertensive medication (e.g., lisinopril/ACE Angiotensin inhibitors ending in "pril", ARB Angiotensin II receptor blockers, spironolactone/Aldactone, Thiazide-type diuretics)

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2027-03-19 (Estimated); Study Completion 2027-03-19 (Estimated)

PRIMARY OUTCOMES:
Diet Adherence | From initiation of ketogenic therapy to the end of treatment (up to 16 weeks)
  The investigators will assess diet adherence primarily by the proportion of youth who maintain an average weekly ketone level of 1 mmol/L or above, as measured through daily blood ketone assays using the Keto Mojo device, a Bluetooth-enabled ketone and glucose testing kit.
Diet Tolerance | From initiation of ketogenic therapy to the end of treatment (up to 16 weeks)
  The investigators will assess diet tolerance primarily by calculating the proportion of youth staying on the diet. The investigators hypothesize 70-80% of youth will tolerate staying on the keto therapy throughout the 16-week treatment as verified by youth self report of continuance of the diet (combined with parent report if applicable). Youth with multiple weekly ketone levels at .5 mmol/L or below will be considered diet intolerant regardless of self-report.
Depression Symptom Improvement | From initiation of ketogenic therapy to the end of treatment (up to 16 weeks)
  The investigators hypothesize that youth who complied with the 16-week keto diet therapy will show statistically significant reductions in depressive symptoms from baseline to completion of the diet. Depressive symptoms will primarily be captured using the clinician-rated Children's Depression Rating Scale, Revised (CDRS-R). Scores range from 17 to 113, with higher scores indicating greater pathology or severity of depressive symptoms (worse outcome).
Bipolar Symptom Improvement | From initiation of ketogenic therapy to the end of treatment (up to 16 weeks)
  The investigators hypothesize that youth who complied with the 16-week keto diet therapy will show statistically significant reductions in bipolar mood instability from baseline to completion of the diet. Bipolar instability will primarily be captured using the clinician-rated Clinical Global Impression - Bipolar Disorder Severity Scale (CGI-BP). CGI-BP overall psychiatric illness scores range from 1 (normal, best outcome) to 7 (very severely ill, worse outcome) and capture severity of bipolar symptoms over the worst 7-day period in the past 2 weeks.
HOMA - IR Metabolic Indicator | From initiation of ketogenic therapy to the end of treatment (up to 16 weeks)
  The investigators hypothesize that youth with high compliance with the keto diet will show significant pre- to post-treatment improvement in Homeostatic model assessment for insulin resistance (HOMA - IR). HOMA - IR is calculated based on fasting glucose and insulin measurements and a value greater than 2 indicates insulin resistance (worse outcome) while a value less than 1 indicates normal range insulin sensitivity (better outcome).

SECONDARY OUTCOMES:
Youth Functional Improvement | From initiation of ketogenic therapy to the end of treatment (up to 16 weeks)
  The investigators hypothesize that youth who complied with the 16-week keto diet therapy will show statistically significant increases in Global Assessment of Functioning (GAF) scores. GAF measures an individual's overall psychological, social, and occupational functioning on a scale from 1 to 100, with higher scores indicating better functioning (better outcome).
Serum Inflammatory Biomarkers (CRP) | From initiation of ketogenic therapy to the end of treatment (up to 16 weeks)
  The investigators hypothesize that youth who complied with the 16-week keto diet therapy will show statistically significant decreases in C-reactive serum protein (CRP) IL-6/IL-10 inflammatory markers. Lower CRP signifies less inflammation (better outcome).

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UCLA Semel Institute Max Gray Child and Adolescent Mood Disorders Program (CHAMP), Los Angeles, California
  - University of Colorado Denver, Anschutz Medical Campus, Aurora, Colorado
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication
Supporting Information: Study Protocol, ICF
Time Frame: 2026-2029
Access Criteria: Researchers may submit a proposal that describes planned analyses to the study PI. Once approved they will be able to access the relevant IPD, protocol and consent documents.

REFERENCES:
- [Background] Yatham LN, Kennedy SH, Parikh SV, Schaffer A, Bond DJ, Frey BN, Sharma V, Goldstein BI, Rej S, Beaulieu S, Alda M, MacQueen G, Milev RV, Ravindran A, O'Donovan C, McIntosh D, Lam RW, Vazquez G, Kapczinski F, McIntyre RS, Kozicky J, Kanba S, Lafer B, Suppes T, Calabrese JR, Vieta E, Malhi G, Post RM, Berk M. Canadian Network for Mood and Anxiety Treatments (CANMAT) and International Society for Bipolar Disorders (ISBD) 2018 guidelines for the management of patients with bipolar disorder. Bipolar Disord. 2018 Mar;20(2):97-170. doi: 10.1111/bdi.12609. Epub 2018 Mar 14. PMID 29536616
- [Background] Wells J, Swaminathan A, Paseka J, Hanson C. Efficacy and Safety of a Ketogenic Diet in Children and Adolescents with Refractory Epilepsy-A Review. Nutrients. 2020 Jun 17;12(6):1809. doi: 10.3390/nu12061809. PMID 32560503
- [Background] Van Meter AR, Burke C, Kowatch RA, Findling RL, Youngstrom EA. Ten-year updated meta-analysis of the clinical characteristics of pediatric mania and hypomania. Bipolar Disord. 2016 Feb;18(1):19-32. doi: 10.1111/bdi.12358. Epub 2016 Jan 9. PMID 26748678
- [Background] Sondike SB, Copperman N, Jacobson MS. Effects of a low-carbohydrate diet on weight loss and cardiovascular risk factor in overweight adolescents. J Pediatr. 2003 Mar;142(3):253-8. doi: 10.1067/mpd.2003.4. PMID 12640371
- [Background] Sondhi V, Agarwala A, Pandey RM, Chakrabarty B, Jauhari P, Lodha R, Toteja GS, Sharma S, Paul VK, Kossoff E, Gulati S. Efficacy of Ketogenic Diet, Modified Atkins Diet, and Low Glycemic Index Therapy Diet Among Children With Drug-Resistant Epilepsy: A Randomized Clinical Trial. JAMA Pediatr. 2020 Oct 1;174(10):944-951. doi: 10.1001/jamapediatrics.2020.2282. PMID 32761191
- [Background] Sethi S, Wakeham D, Ketter T, Hooshmand F, Bjornstad J, Richards B, Westman E, Krauss RM, Saslow L. Ketogenic Diet Intervention on Metabolic and Psychiatric Health in Bipolar and Schizophrenia: A Pilot Trial. Psychiatry Res. 2024 May;335:115866. doi: 10.1016/j.psychres.2024.115866. Epub 2024 Mar 20. PMID 38547601
- [Background] Miklowitz DJ, Schneck CD, Walshaw PD, Singh MK, Sullivan AE, Suddath RL, Forgey Borlik M, Sugar CA, Chang KD. Effects of Family-Focused Therapy vs Enhanced Usual Care for Symptomatic Youths at High Risk for Bipolar Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2020 May 1;77(5):455-463. doi: 10.1001/jamapsychiatry.2019.4520. PMID 31940011
- [Background] Miklowitz DJ, Schneck CD, George EL, Taylor DO, Sugar CA, Birmaher B, Kowatch RA, DelBello MP, Axelson DA. Pharmacotherapy and family-focused treatment for adolescents with bipolar I and II disorders: a 2-year randomized trial. Am J Psychiatry. 2014 Jun;171(6):658-67. doi: 10.1176/appi.ajp.2014.13081130. PMID 24626789
- [Background] Kossoff EH, Zupec-Kania BA, Auvin S, Ballaban-Gil KR, Christina Bergqvist AG, Blackford R, Buchhalter JR, Caraballo RH, Cross JH, Dahlin MG, Donner EJ, Guzel O, Jehle RS, Klepper J, Kang HC, Lambrechts DA, Liu YMC, Nathan JK, Nordli DR Jr, Pfeifer HH, Rho JM, Scheffer IE, Sharma S, Stafstrom CE, Thiele EA, Turner Z, Vaccarezza MM, van der Louw EJTM, Veggiotti P, Wheless JW, Wirrell EC; Charlie Foundation; Matthew's Friends; Practice Committee of the Child Neurology Society. Optimal clinical management of children receiving dietary therapies for epilepsy: Updated recommendations of the International Ketogenic Diet Study Group. Epilepsia Open. 2018 May 21;3(2):175-192. doi: 10.1002/epi4.12225. eCollection 2018 Jun. PMID 29881797
- [Background] Ildarabadi A, Mir Mohammad Ali SN, Rahmani F, Mosavari N, Pourbakhtyaran E, Rezaei N. Inflammation and oxidative stress in epileptic children: from molecular mechanisms to clinical application of ketogenic diet. Rev Neurosci. 2024 Feb 14;35(4):473-488. doi: 10.1515/revneuro-2023-0128. Print 2024 Jun 25. PMID 38347675
- [Background] Gundogdu U, Gurer G, Eroglu M. Executive function, behavioral problems, and insulin resistance in adolescents with obesity. J Pediatr Endocrinol Metab. 2023 Apr 19;36(6):539-546. doi: 10.1515/jpem-2022-0510. Print 2023 Jun 27. PMID 37071665
- [Background] Goldstein BI, Birmaher B, Carlson GA, DelBello MP, Findling RL, Fristad M, Kowatch RA, Miklowitz DJ, Nery FG, Perez-Algorta G, Van Meter A, Zeni CP, Correll CU, Kim HW, Wozniak J, Chang KD, Hillegers M, Youngstrom EA. The International Society for Bipolar Disorders Task Force report on pediatric bipolar disorder: Knowledge to date and directions for future research. Bipolar Disord. 2017 Nov;19(7):524-543. doi: 10.1111/bdi.12556. Epub 2017 Sep 25. PMID 28944987
- [Background] Dsouza A, Haque S, Aggarwal R. The influence of ketogenic diets on mood stability in bipolar disorder. Asian J Psychiatr. 2019 Mar;41:86-87. doi: 10.1016/j.ajp.2017.10.024. Epub 2017 Oct 28. No abstract available. PMID 29169915
- [Background] Batt, M., Miklowitz, D. J., Elliotte, E., Hafeman, D., Birmaher, B., Delbello, M. P., Stepanova, E., Findling, R., Goldstein, B, I., Post, R., & Schneck, C. D. (2024). A survey of expert psychiatrists regarding first- and second-line medication choices for pediatric bipolar disorder. Bipolar Disorders, 26, 119.
- See also: UCLA Child Bipolar Network Research Studies Page — https://www.semel.ucla.edu/champ/max-gray-champ-research
- See also: Study info: U of Colorado Denver - Anschutz Medical Campus — https://researchstudies.cuanschutz.edu/Study/24-2497